CLINICAL TRIAL: NCT04521101
Title: Can we Make a VAST Improvement? Promoting Anaesthetists' Non-technical Skills Through the Vital Anaesthesia Simulation Training Course in a Low-resource Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Patricia Livingston, Professor, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-4474
Record Dates: First submitted 2019-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: To Determine the Change in Demonstrated Anesthesia Non-technical Skills After Delivery of the VAST Course

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VAST Course (Other)
  Interventions: Other: VAST Course

INTERVENTIONS:
Other: VAST Course — Educational course to teach non-technical skills

SUMMARY:
Rationale: The World Health Assembly resolution 68.15 identified surgical and anesthesia care as core components of universal health coverage. However, about 5 billion people worldwide lack access to essential surgical and anesthesia services. Of the 313 million procedures undertaken each year only 6% occur in the poorest countries with an estimated 30% of all deaths globally associated with common surgical conditions. Patient safety in low-resource settings is hindered by severe workforce shortages, lack of essential resources, hierarchical culture and few opportunities for professional development.

Non-technical skills (NTS), such as communication, team working, and task coordination, are vital to patient safety. Up to 70-80% of untoward events in health care are associated with errors in NTS8. The Anaesthetists' Non-Technical Skills framework (ANTS) describes behaviour markers for NTS in anesthesia. This framework has been found applicable in low-resource settings.

Simulation-based education is widespread for NTS training in well-resourced countries. Traditionally, high costs have prohibited this modality in low-resource settings. Foundational work in Rwanda and at Dalhousie University has demonstrated that effective training in ANTS can be achieved through simple low-cost simulation. The Vital Anaesthesia Simulation Training (VAST) Course is a three-day simulation-based program designed de-novo to focus on core clinical practices and NTS that promote safe perioperative care in low-resource settings. The course uses low-cost materials in an immersive simulated environment to replicate common cases managed in district hospitals in low-resource settings. Realism is created with simple mannequins, iPads with the SimMon App functioning as monitoring, basic props (e.g., airway equipment, syringes, drapes), photographs of pathology, and briefing cards for scenario role-play.

Purpose: To assess the impact of the VAST Course on ANTS and explore factors that influence long-term retention of ANTS amongst anesthesia providers in a low-resource setting.

ELIGIBILITY:
Inclusion Criteria:

* All anesthesia (anesthesiologists, anesthesia residents and non-physician anesthetists) VAST Course participants during the study period.

Exclusion Criteria:

* VAST Course participants who do not practice anesthesia (surgeons, nurses, midwives etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Total Anesthesia NonTechnical Skills (ANTS) Score | Day 1 (pre-course test)
  Baseline ANTS Score
Total Anesthesia NonTechnical Skills (ANTS) Score | Day 3 (post-course test)
  The change from baseline ANTS score to post-course (day 3)
Total Anesthesia NonTechnical Skills (ANTS) Score | 4 months (follow-up score)
  The change from baseline ANTS score to follow-up (4 months)

SECONDARY OUTCOMES:
Category Anesthesia NonTechnical Skills (ANTS) Score | Day 1 (pre-course)
  Baseline category ANTS scores (team working, task management, situation awareness, decision making)
Category Anesthesia NonTechnical Skills (ANTS) Score | Day 3 (post-course)
  The change in category ANTS scores (team working, task management, situation awareness, decision making)
Category Anesthesia NonTechnical Skills (ANTS) Score | 4 months (post-course)
  The change in category ANTS scores (team working, task management, situation awareness, decision making)

CONTACTS AND LOCATIONS:
Locations (2):
- Rwanda (2):
  - University of Rwanda, Butare
  - Rwanda Military Hospital, Kigali

IPD SHARING:
Plan to Share IPD: No